CLINICAL TRIAL: NCT01613482
Title: Interest of the Prophylactic Cerebral Radiotherapy in the Metastatic Breast Cancer Expressing HER2/NEU Treated by Trastuzumab
Brief Title: TraStuzumAb-Radiotherapy : Impact on the Cerebral Prevention
Acronym: TSARINE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSARINE 0602
Record Dates: First submitted 2012-06-01; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer; Metastasis; Sur-expressing Her2-neu
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Without cerebral prophylactic radiation
  Interventions: Drug: Trastuzumab; Drug: Other chemotherapy in association with Trastuzumab
- Arm B (Experimental): With cerebral prophylactic radiation
  Interventions: Radiation: cerebral prophylactic radiation; Drug: Trastuzumab; Drug: Other chemotherapy in association with Trastuzumab

INTERVENTIONS:
Radiation: cerebral prophylactic radiation — 24Gy, 12 fractions of 2 Gy
  Arms: Arm B
Drug: Trastuzumab — Weekly, 2mg/kg of corporal weight
Drug: Other chemotherapy in association with Trastuzumab — other chemotherapy is possible to associate with Trastuzumab as well as a change of chemotherapy protocol is possible while maintening Trastuzumab 8 weeks is required between last injection of chemotherapy and first radiotherapy session

SUMMARY:
Evaluate the survival without metastasis in patients treated by Trastuzumab in association with other chemotherapies for a breast cancer expressing HER2-NEU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer, expressing HER2-NEU (score +++ in ICH or ++ and amplification on FISH or CISH, SISH)
* Visceral metastasis, only or multiple
* First line metastasis treatment by Trastuzumab in association with chemotherapy
* Good general conditions: OMS=<2 or Karnofsky >=70%
* Age > 18 years and < 70 years
* Life expectancy >=3 mois
* No Trastuzumab since more of 6 months
* No cerebral metastasis (MRI)
* Efficacy contraception for women with genital capacities
* Consent signed by the patient

Exclusion Criteria

* Contraindication to IRM
* Psychiatric decease
* Prior cerebral radiotherapy,
* Geographical constraint, compromising the fallow of patients
* Infectious or other serious pathology, likely to stop the treatment
* Positive serology (HIV, hBC, hBS)
* Inclusion in an other clinical trial or in the 4 weeks before th inclusion
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
free of cerebral metastasis survival | 5 years

SECONDARY OUTCOMES:
survival (overall and free visceral progression) | 5 years
evaluate neurological, haemorrhagic, skin toxicities | During study
  weekly during radiotherapy and 2 weeks after radiotherapy
neurological toxicities | During study
  * neurological exams
  * Cognitive test
  * Subjective questionnaire of cognitive complaint
  * questionnaire of EORTC QLQ-BN20
P105 value | prior to trastuzumab, after 3 months, 6 months, 12 months, 18 months, 24 months, 36 months
  Blood sample
quality of life | before treatment, after 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Questionnaire QLQ-bn20

CONTACTS AND LOCATIONS:
Overall Officials: Yazid BELKACEMI, MD, Principal Investigator — y-belkacemi@o-lambret.fr
Locations (26):
- France (26):
  - Centre Paul Papin, Angers
  - Centre Hospitalier, Boulogne-sur-Mer
  - Centre Maurice Tubiana, Caen
  - Centre G-François Baclesse, Caen
  - Centre Léonard de Vinci, Dechy
  - Centre Médical de Forcilles, Forcilles-attilly
  - Clinique des Ormeaux- Vauban, Le Havre
  - Centre Bourgogne, Lille
  - Centre Oscar LAMBRET, Lille
  - CHU Dupuytren, Limoges
  - Clinique Clinique Clementville, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Catherine de Sienne, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Centre médical Oncogard, Nîmes
  - Hôpital Tenon, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier LYON SUD, Pierre-Bénite
  - Centre René Huguenin, Saint-Cloud
  - Centre Etienne DOLET, Saint-Nazaire
  - Centre de Cancérologie Paris Nord, Sarcelles
  - Oncorad Garonne, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif